CLINICAL TRIAL: NCT06260800
Title: Translation, Adaptation and Valitation of the Spanish Version of Credibility and Expectancy Questionnaire in Patiens With Musculoskeletal Injuries
Brief Title: Spanish Version of Credibility and Expectancy Questionnaire in Patients With Musculoskeletal Injuries
Status: Completed | Type: Observational
Sponsor: University of Valladolid (Other)
Responsible Party: Principal Investigator, Silvia Lahuerta Martín, Principal investigator, University of Valladolid
Other Study IDs: PI 23-3405
Record Dates: First submitted 2023-12-18; First posted 2024-02-15 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2024-12

CONDITIONS: Validation Study

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CEQ Validation: In initial assessment, EQ-5D-5L and HADS questionnaires were completed. After sessions 1 and 2, CEQ and WAI-S were filled. Finally, EQ-5D-5L was completed before the fourth session.
  Interventions: Other: Validation CEQ

INTERVENTIONS:
Other: Validation CEQ — In initial assessment, EQ-5D-5L and HADS questionnaires were completed. After sessions 1 and 2, CEQ and WAI-S were filled. Finally, EQ-5D-5L was completed before the fourth session.

SUMMARY:
Physiotherapy treatment of musculoskeletal injuries should be performed following the main clinical guidelines of person-centered care. Patients' perception of the abilities and facilities provided by physiotherapists boost a convenient therapeutic relationship. This relation is linked with more satisfaction and adherence during the treatment, as well as credibility and expectancy of the patient related to the treatment. Thus, Credibility and Expectancy questionnaire is normally used to assess that point. CEQ presents good psychometric properties when used in Physisiotherapy interventions, but there is not a spanish version of this questionaire.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer patients who are going to start physiotherapy treatment due to musculoskeletal injuries.
* Age above 18 years old.
* Understanding of the study purpose and signing the informed consent.

Exclusion Criteria:

* Patients with cognitive deprivation.
* Not able to fill in the questionnaires autonomously.
* Mother tongue different from Spanish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are going to start physiotherapy treatment due to musculoskeletal injuries.
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Content validity | During the intervention: Session 1
  Credibility and Expectancy questionnaire (CEQ) must be completed, while registering the time used and the quality and the reading comprehension.
Structural validity | During the intervention: session 1 and 2 treatment
  Exploratory factor analysis (EFA) and confirmatory factorial analysis (CFA) were performed. For EFA Kaiser criterion >0.70 will be acceptable. For CFA, goodness of fit index and comparative fit index were calculated, where values up to 0.90 were acceptable.
Reliability | During the intervention.
  Credibility and Expectancy questionnaire (CEQ) reliability will be analised through internal consistency (alpha Cronbach > 0.70 recomended)) and test-retest (intraclass correlation coeficient >0.70 acceptable).
Hypotheses testing for construct validity | During the intervention.
  Comparing CEQ with other measurement instruments.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Lahuerta Martín, Principal Investigator — University of Valladolid, Soria, Spain
Locations (1):
- Silvia Lahuerta Martín, Soria, Spain

IPD SHARING:
Plan to Share IPD: No